CLINICAL TRIAL: NCT00375531
Title: Use of Mindfulness Meditation With Iraqi/Afghanistan War Veterans With Post Traumatic Stress Disorder
Brief Title: Use of Mindfulness Meditation With Iraqi/Afghanistan War Veterans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol revisions were deemed unable to be completed by 8/2007
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other); University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00890; USUHS #PA181BO-4
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2007-10

CONDITIONS: PTSD; Stress
Keywords: Post Traumatic Stress Disorder; Mindfulness Meditation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness Meditation (MfM)

SUMMARY:
Objectives: The primary objective of this study is to conduct a randomized pilot study on the efficacy of Mindfulness Meditation (MfM) on sleep in post war Iraqi/Afghanistan veterans with PTSD. It is hypothesized that the change in sleep (measured by actigraphy), sleep self report measures, and PTSD symptoms (measured by the PTSD Checklist) from baseline, 8 weeks and 12 weeks will be greater for veterans with PTSD who are treated with MfM, controlling for pretreatment values and other clinical and demographic factors.

A secondary objective will investigate whether there is an improvement in psychological wellness (measured by optimism, perceived wellness, and spirituality) following MfM treatments.

It is hypothesized that change in optimism, perceived wellness, and spirituality from baseline, 8 weeks and 12 weeks will improve in veterans with PTSD who are treated with MfM, controlling for pretreatment values and other clinical and demographic factors. Physiological measures of actigraphy in the home will be done at baseline, eight weeks, and twelve weeks. Subjective measure of sleep include measurements of sleep and quality of life(FOSQ) and subjective sleep quality (PSQI). Other self-report measures that will examine psychological wellness include the Life Orientation Test (LOT), the Perceived Wellness Survey (PWS) and the Spirituality Assessment Scale (SAS).

DETAILED DESCRIPTION:
Research Design: This exploratory study is a randomized, controlled, repeated measures trial to estimate the effectiveness of mindfulness meditation (MfM) to improve the severity of PTSD symptoms, specifically sleep and anxiety, and to improve the psychological wellbeing in Iraqi veterans with PTSD. The study is a repeated measures, comparative study using a parallel design. Both groups will receive routine treatment for PTSD; in addition, the treatment group will receive 8 weeks (1.5 hours/week) of mindfulness meditation from a trained psychologist, (Co-PI, N Chychula) who has been conducting these mindfulness meditation groups with combat veterans for 3 years. Subjects will be asked to commit to practice mindfulness meditation practice for 45 minutes each day. Data will be collected at baseline, eight weeks, and twelve weeks (one month follow-up). An equal number of participants will be randomly assigned to each group with 15 assigned to each group.

Methodology: For purposes of this pilot study, mindfulness meditation will be delivered in the context of a structured manual driven program, developed to enhance awareness of moment-to-moment experience of perceived mental processes. Although rooted in Buddhist traditions, this program is not religious but aims to create a greater awareness of body sensations, feelings and thoughts. This is thought to allow greater perception of one's responses and a gradual reduction in negative affect accompanied by an improvement in vitality and coping and psychological wellbeing (Grossman, 2004).

ELIGIBILITY:
INCLUSION CRITERIA:

* Iraqi War veterans who have returned from deployment for at least 3 months
* The veterans must be willing to practice MfM for 45 minutes each day and agree to follow all treatment protocols.

EXCLUSION CRITERIA:

Patients with a documented diagnosis of:

* a thought disorder
* a bipolar disorder
* a borderline personality disorder
* active substance abuse/dependence,

Patients that are:

* homeless
* have pending legal dispositions
* are unable to hear, read, visualize, and/or comprehend the assessment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Sleep & PTSD SYMPTOM SEVERITY -- (measured by) Actigraphy, PTSD Checklist (PCL), Functional Outcomes of Sleep Questionnaire (FOSQ),Pittsburgh Sleep Quality Index (PSQI) -- Self-report measures and actigraphy readings will be
collected at baseline, 8 weeks, and 12 weeks in
both groups.

SECONDARY OUTCOMES:
PSYCHOLOGICAL WELLNESS ASSESSMENTS -- (measured by) Life Orientation Test (LOT), Perceived Wellness Survey (PWS), Spirituality Assessment Scale (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Nina M Chychula, Ph.D., Principal Investigator — Philadelphia VAMC and University of Pennsylvania
Locations (1):
- Philadelphia VAMC, Philadelphia, Pennsylvania, United States